CLINICAL TRIAL: NCT03556592
Title: An Open-label, Multi Centre Drug-drug Interaction Trial to Investigate the Effects of Tralokinumab on the Pharmacokinetics of Selected Cytochrome P450 Substrates in Adult Subjects With Moderate-to-severe Atopic Dermatitis
Brief Title: Drug-drug Interaction Trial With Tralokinumab in Moderate to Severe Atopic Dermatitis - ECZTRA 4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP0162-1342; 2018-000534-35 (EudraCT Number)
Record Dates: First submitted 2018-05-30; First posted 2018-06-14 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2020-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tralokinumab; Caffeine; Warfarin; Omeprazole; Metoprolol; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): Tralokinumab - investigational medicinal product:
  Week 0: subcutaneous (SC) injection of tralokinumab loading dose.
  Week 2 to Week 14: SC injection of tralokinumab maintenance dose.
  CYP substrates - non-investigational medicinal products:
  Week -1, Week 1, and Week 15: oral administration of caffeine 100 mg, warfarin sodium 5 mg x2, omeprazole 20 mg, metoprolol tartrate 100 mg, and midazolam hydrochloride 2 mg.
  Interventions: Drug: Tralokinumab; Drug: Caffeine; Drug: Warfarin; Drug: Omeprazole; Drug: Metoprolol; Drug: Midazolam Hydrochloride

INTERVENTIONS:
Drug: Tralokinumab — Human recombinant monoclonal antibody of the IgG4 subclass that specifically binds to human IL-13 and blocks interaction with the IL-13 receptors. Presented as a liquid formulation for subcutaneous injection.
Drug: Caffeine — 1x 100 mg tablet
Drug: Warfarin — 2x 5 mg tablets
Drug: Omeprazole — 1x 20 mg capsule
Drug: Metoprolol — 1x 100 mg tablet
Drug: Midazolam Hydrochloride — 1 mL of 2 mg/mL oral solution/syrup

SUMMARY:
The purpose of this trial is to investigate if tralokinumab changes the metabolism of selected CYP substrates in adults with moderate-to-severe AD after:

* 14 weeks of treatment with tralokinumab
* a single dose of tralokinumab

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above.
* Diagnosis of AD as defined by the Hanifin and Rajka 1980 criteria for AD.
* History of AD for ≥1 year.
* Subjects who have a recent history of inadequate response to treatment with topical medications or for whom topical treatments are otherwise medically inadvisable.
* AD involvement of ≥10% body surface area at screening and baseline.
* Stable dose of emollient twice daily (or more, as needed) for at least 14 days before baseline.
* Willingness to abstain from consumption of any 1 or more of the following items in the periods specified:

  * ±7 days within each cocktail dosing visit: foods/beverages that affect the CYP system:

    * Grapefruit or grapefruit juice, Seville oranges or orange juice, starfruit, pomegranate and cranberry juices, red wine, red grape extract.
    * Cruciferous vegetables (for example broccoli).
    * Chargrilled meat.
  * ±48 hours within each cocktail dosing visit: caffeinated beverages and foods/drugs that contain caffeine.

Exclusion Criteria:

* Administration, within 14 days or 5 half-lives (whichever is longer) prior to Day -7, of any medication that is a known inducer or inhibitor of 1 or more of the following CYP enzymes: CYP3A, CYP2C19, CYP2C9, CYD2D6, and CYP1A2.
* Subjects who are poor metabolisers of CYP2C9, CYP2C19, or CYP2D6, based on genotyping.
* Any contraindication to 1 or more of the following drugs, according to the applicable labelling: caffeine, warfarin, omeprazole, metoprolol, or midazolam.
* Consumption of any 1 or more of the following items in the periods specified:

  * ±7 days within each cocktail dosing visit: foods/beverages that affect the CYP system:

    * Grapefruit or grapefruit juice, Seville oranges or orange juice, starfruit, pomegranate and cranberry juices, red wine, red grape extract.
    * Cruciferous vegetables (for example broccoli).
    * Chargrilled meat.
  * ±48 hours within each cocktail dosing visit: caffeinated beverages and foods/drugs that contain caffeine.
* Nausea or diarrhoea 1 week prior to Day -7.
* Active dermatologic conditions that may confound the diagnosis of AD.
* Use of tanning beds or phototherapy within 5 weeks prior to Day -7.
* Treatment with systemic immunosuppressive/immunomodulating drugs and/or systemic corticosteroid within 3 weeks prior to Day -7.
* Treatment with topical corticosteroids, topical calcineurin inhibitors, or topical phosphodiesterase 4 inhibitors within 1 week prior to Day -7.
* Receipt of any marketed biological therapy or investigational biologic agent (including immunoglobulin, anti-IgE, or dupilumab):

  * Any cell-depleting agents, including but not limited to rituximab: within 6 months prior to Day -7, or until lymphocyte count returns to normal, whichever is longer.
  * Other biologics: within 3 months or 5 half-lives, whichever is longer, prior to Day -7.
* Active skin infection within 1 week prior to Day -7.
* Clinically significant infection within 4 weeks prior to Day -7.
* A helminth parasitic infection within 6 months prior to the date informed consent is obtained.
* Tuberculosis requiring treatment within 12 months prior to screening.
* Known primary immunodeficiency disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Ratio of the AUC-last at Week 15 (after multiple doses of tralokinumab) to that on Day -7 (at baseline) for each of the 5 substrates | Day -7 and Week 15
  AUC-last = area under the plasma concentration curve from time 0 to the last quantifiable observation
Ratio of the Cmax at Week 15 (after multiple doses of tralokinumab) to that on Day -7 (at baseline) for each of the 5 substrates | Day -7 and Week 15
  Cmax = maximum observed plasma concentration

SECONDARY OUTCOMES:
Ratio of the AUC-last on Day 8 (after a single dose of tralokinumab) to that on Day -7 (at baseline) for each of the 5 substrates | Day -7 and Day 8
  AUC-last = area under the plasma concentration curve from time 0 to the last quantifiable observation
Ratio of the Cmax on Day 8 (after a single dose of tralokinumab) to that on Day -7 (at baseline) for each of the 5 substrates | Day -7 and Day 8
  Cmax = maximum observed plasma concentration
Ratio of the AUC-inf on Day 8 (after a single dose of tralokinumab) to that on Day -7 (at baseline) for each of the 5 substrates | Day -7 and Day 8
  AUC-inf = area under the plasma concentration curve from time 0 to infinity
Number of adverse events | From Day 1 up to Week 30
Presence of anti-drug antibodies (yes/no) | From Day 1 up to Week 30

CONTACTS AND LOCATIONS:
Overall Officials: Medical expert, Study Director — LEO Pharma
Locations (11):
- United States (8):
  - LEO Pharma Investigational Site, Little Rock, Arkansas
  - LEO Pharma Investigational Site, Rogers, Arkansas
  - LEO Pharma Investigational Site, San Diego, California
  - LEO Pharma Investigational Site, Doral, Florida
  - LEO Pharma Investigational Site, Miami, Florida
  - LEO Pharma Investigational Site, Quincy, Massachusetts
  - LEO Pharma Investigational Site, Spartanburg, South Carolina
  - LEO Pharma Investigational Site, Norfolk, Virginia
- France (2):
  - LEO Pharma Investigational Site, Nice
  - LEO Pharma Investigational Site, Paris
- LEO Pharma Investigational Site, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No